CLINICAL TRIAL: NCT04592198
Title: A Randomized, Dose-ranging, Open-label, Parallel Group Study to Assess the Efficacy, Safety and Pharmacokinetics of Palonosetron HCl Buccal Film Versus IV Palonosetron 0.25 mg for the Prevention of CINV in Cancer Patients Receiving MEC
Brief Title: Buccal Film Versus IV Injection Palonosetron for Moderately Emetogenic Chemotherapy Induced Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xiamen LP Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LP-CT-PALO-202002
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Nausea With Vomiting Chemotherapy-Induced
MeSH Terms: interventions — Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A (Buccal 0.25 Mg) (Experimental): Palonosetron HCl Buccal Film 0.25 Mg
  Interventions: Drug: Palonosetron Hydrochloride Buccal Film 0.25 Mg
- B (Buccal 0.5 Mg) (Experimental): Palonosetron HCl Buccal Film 0.5 Mg
  Interventions: Drug: Palonosetron Hydrochloride Buccal Film 0.5 Mg
- C (IV Injection 0.25 Mg) (Active Comparator): IV palonosetron 0.25 Mg (ALOXI®)
  Interventions: Drug: Palonosetron Hydrochloride, 0.25 Mg/5 mL Intravenous Solution

INTERVENTIONS:
Drug: Palonosetron Hydrochloride Buccal Film 0.25 Mg — Dose equal to the iv control
  Other Names: Buccal Film Low Dose
  Arms: A (Buccal 0.25 Mg)
Drug: Palonosetron Hydrochloride Buccal Film 0.5 Mg — Dose twice that of iv control
  Other Names: Buccal Film High dose
  Arms: B (Buccal 0.5 Mg)
Drug: Palonosetron Hydrochloride, 0.25 Mg/5 mL Intravenous Solution — iv control
  Other Names: Control Standard Treatment (Aloxi)
  Arms: C (IV Injection 0.25 Mg)

SUMMARY:
Phase 2 study to compare efficacy, safety and PK of palonosetron, a long acting 5-HT3 receptor antagonist, by buccal film delivery compared to iv injection for chemotherapy induced nausea or vomiting (CINV). Subjects receive a single dose of palonosetron prior to moderately emetogenic chemotherapy.

DETAILED DESCRIPTION:
This is a Phase 2 study to compare efficacy, safety and PK of palonosetron, a long acting 5-HT3 receptor antagonist, by buccal film compared to iv injection for moderately emetogenic chemotherapy-induced nausea or vomiting (CINV) in cancer patients. Subjects are randomized into three treatment groups, two with the experimental study drug palonosetron in buccal film at one of two different doses or the control treatment using Palonosetron hydrochloride iv injection. Palonosetron PK will be assessed in a subgroup of each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* With histologically or cytologically confirmed malignant disease;

  -. Be scheduled to receive the first course of MEC to be administered on Day 1
* Using reliable contraceptive measures;
* negative serum pregnancy test (if potentially child bearing)

Exclusion Criteria:

* Received investigational drugs within 30 days before the start of study treatment or scheduled to receive a highly or moderately emetogenic chemotherapeutic agent;
* Have a clinically unstable seizure disorder with seizure activity requiring anticonvulsant medication;
* Have severe renal or hepatic impairment;
* Have positive serology test results;
* Have a known contraindication to 5-HT3 receptor antagonists;
* Treated with commercially available or investigative palonosetron formulation within 2 weeks prior to start of study treatment;
* Allergic to palonosetron or any other 5-HT3 antagonist;
* Currently a user of any recreational or illicit drugs (including marijuana) or has current evidence of drug or alcohol abuse or dependence as determined by the investigator;
* Will be receiving stem cell rescue therapy in conjunction with study related course of emetogenic chemotherapy;
* Received or will receive total body irradiation or radiation therapy to the abdomen or pelvis in the week prior to Treatment Day 1 and/or during the diary reporting period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjit Nirmalanandhan, Ph.D., Principal Investigator — Ocala Oncology Center PL DBA Florida Cancer Affiliates
Locations (7):
- United States (7):
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - Ocala Oncology Center PL DBA Florida Cancer Affiliates, Ocala, Florida
  - Edward H. Kaplan MD & Associates, Skokie, Illinois
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Monongahela Valley Hospital/ Regional Cancer Center, Monongahela, Pennsylvania
  - Charleston Oncology, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A (Buccal 0.25 Mg) | B (Buccal 0.5 Mg) | C (IV Injection 0.25 Mg)
Started | 8 | 8 | 6
Completed | 7 | 8 | 6
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject in Group A withdrew consent and was withdrawn (no additional information was provided).
Groups:
- Total: Total of all reporting groups
Arm/Group | A (Buccal 0.25 Mg) | B (Buccal 0.5 Mg) | C (IV Injection 0.25 Mg) | Total
Number analyzed (Participants) | 7 | 8 | 6 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (9.32) | 53.9 (10.96) | 59.8 (9.13) | 58.8 (10.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 6 | 16
  Male | 2 | 3 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 5 | 8 | 4 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
History of motion sickness [Number; unit: participants]
  Yes | 1 | 2 | 1 | 4
  No | 6 | 6 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Complete Acute Response
Description: no emetic episode and no rescue medication during the first 24 hours after chemotherapy
Time Frame: first 24 hours after chemotherapy
Measure: Count of Participants; unit: Participants
Groups:
- B (Buccal 0.50 Mg): Palonosetron HCl Buccal Film 0.5 Mg
- C (IV Injection 0.25 Mg): IV palonosetron 0.25 Mg (ALOXI)
Arm/Group | A (Buccal 0.25 Mg) | B (Buccal 0.50 Mg) | C (IV Injection 0.25 Mg)
Number analyzed (Participants) | 7 | 8 | 5
Participants | 4 | 4 | 3

ADVERSE EVENTS:
Time Frame: Adverse event reporting begins from the time of informed consent to the end of that last visit (Visit 5, Day 9 (for non-PK group)/ Day 11 (for PK group)).
Description: All subjects in the safety population received the planned single dose of study drug: Palonosetron HCl Buccal Film 0.25mg for 7 subjects, Palonosetron HCl Buccal Film 0.5 mg for 8 subjects, and ALOXI® for 6 subjects
Groups:
- C (IV Injection 0.25Mg): IV palonosetron 0.25 Mg (ALOXI®)
Arm/Group | A (Buccal 0.25 Mg) | B (Buccal 0.5 Mg) | C (IV Injection 0.25Mg)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT04592198/Prot_SAP_001.pdf